CLINICAL TRIAL: NCT01970371
Title: A Phase 3, Multicenter, Randomized, Open-Label Study to Evaluate the Efficacy and Safety of Plazomicin Compared With Colistin in Patients With Infection Due to Carbapenem-Resistant Enterobacteriaceae (CRE)
Brief Title: A Study of Plazomicin Compared With Colistin in Patients With Infection Due to Carbapenem-Resistant Enterobacteriaceae (CRE)
Acronym: CARE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Achaogen, Inc. (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACHN-490-007; 2013-001997-18 (EudraCT Number); U1111-1151-2686 (Other: WHO)
Record Dates: First submitted 2013-10-23; First posted 2013-10-28 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Bloodstream Infections (BSI) Due to CRE; Hospital-Acquired Bacterial Pneumonia (HABP) Due to CRE; Ventilator-Associated Bacterial Pneumonia (VABP) Due to CRE; Complicated Urinary Tract Infection (cUTI) Due to CRE; Acute Pyelonephritis (AP) Due to CRE
Keywords: Gram-negative; bacterial infection; antibacterial; antimicrobial; CRE; CPE; BSI; pneumonia; HABP; VABP; AP; cUTI; UTI
MeSH Terms: conditions — Sepsis; Bacterial Infections; Pneumonia | interventions — plazomicin; Colistin; colistinmethanesulfonic acid; Meropenem; Tigecycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Plazomicin in Combination with Meropenem or Tigecycline (Experimental): Cohort 1: Patients received 15 milligram per killogram (mg/kg) plazomicin therapy (plus meropenem or tigecycline) as a 30-minute intravenous (IV) infusion once daily for 7 to 14 days.
  Interventions: Drug: plazomicin; Drug: meropenem; Drug: tigecycline
- Colistin in Combination with Meropenem or Tigecycline (Active Comparator): Cohort 1: Patients received a 5 mg/kg IV loading dose (300 mg maximum) colistin (plus meropenem or tigecycline) followed by a 5 mg/kg/d maintenance dose divided into every 8 hours (q8h) or every 12 hours (q12h) for 7 to 14 days.
  Interventions: Drug: colistin; Drug: meropenem; Drug: tigecycline
- Plazomicin in Combination with Adjunctive Antibiotic (Experimental): Cohort 2: Patients received 15 mg/kg as a 30 minute IV infusion once daily. BSI, HABP or VABP patients received plazomicin and any supplemental antibiotic therapy, according to Investigator's choice, for 7 to 14 days. cUTI or AP patients received plazomicin monotherapy only for 4 to 7 days with an option to switch to oral therapy on or after Day 5.
  Interventions: Drug: plazomicin; Drug: antibiotic of Investigator's choice

INTERVENTIONS:
Drug: plazomicin
  Arms: Plazomicin in Combination with Adjunctive Antibiotic; Plazomicin in Combination with Meropenem or Tigecycline
Drug: colistin
  Other Names: colistimethate sodium
  Arms: Colistin in Combination with Meropenem or Tigecycline
Drug: meropenem
  Arms: Colistin in Combination with Meropenem or Tigecycline; Plazomicin in Combination with Meropenem or Tigecycline
Drug: tigecycline
  Arms: Colistin in Combination with Meropenem or Tigecycline; Plazomicin in Combination with Meropenem or Tigecycline
Drug: antibiotic of Investigator's choice
  Arms: Plazomicin in Combination with Adjunctive Antibiotic

SUMMARY:
This was a Phase 3 study containing a randomized open-label superiority cohort (Cohort 1) comparing the efficacy and safety of plazomicin with colistin when combined with a second antibiotic (either meropenem or tigecycline) in the treatment of patients with bloodstream infection (BSI), hospital acquired bacterial pneumonia (HABP), or ventilator-associated bacterial pneumonia (VABP) due to CRE. An additional cohort of patients with BSI, HABP, VABP, complicated urinary tract infection (cUTI), or acute pyelonephritis (AP) due to CRE, not eligible for inclusion in the other cohort, were enrolled into a single arm (Cohort 2) and treated with plazomicin-based therapy. Therapeutic drug management (TDM) was used to help ensure that plazomicin exposures lie within an acceptable range of the target mean steady-state area under the curve (AUC).

ELIGIBILITY:
Key Inclusion Criteria:

* Cohort 1: APACHE II score between 15 and 30, inclusive; Cohort 2: BSI, HABP, VABP patients with an APACHE II score ≤30 (cUTI and AP patients do not need to have their APACHE II score calculated)
* Positive culture that was collected ≤96 hours prior to randomization indicating a CRE infection, or a high likelihood of a CRE infection
* Diagnosis of BSI as defined by at least one of the following: fever, hypothermia, new onset arterial hypotension, elevated total peripheral white blood cell (WBC) count, increased immature neutrophils (band forms), or leukopenia
* Or, diagnosis of HABP defined as clinical signs and symptoms consistent with pneumonia acquired after at least 48 hours of continuous stay in an inpatient acute or chronic-care facility, or acquired within 7 days after being discharged from a hospitalization of ≥3 days duration
* Or, diagnosis of VABP defined by clinical signs and symptoms consistent with pneumonia acquired after at least 48 hours of continuous mechanical ventilation
* Or, diagnosis of cUTI or AP defined by clinical signs and symptoms consistent with cUTI or AP assessed within 24 hours prior to enrollment

Key Exclusion Criteria:

* Cohorts 1 and 2 BSI, HABP, and VABP patients: receipt of more than 72 hours of potentially effective antibacterial therapy; Cohort 2: cUTI and AP patients: receipt of any potentially effective antibacterial therapy in the 48 hours prior to enrollment
* Cohort 1 only: knowledge that index CRE infection is resistant to colistin prior to randomization
* Objective clinical evidence for any of the following clinical syndromes that necessitates study therapy for greater than 14 days: endovascular infection including endocarditis, osteomyelitis, prosthetic joint infection, meningitis and/or other central nervous system infections
* Objective clinical evidence of infectious involvement of intravascular material potentially due to the study qualifying pathogen and not intended to be removed within 4 calendar days of the initial positive culture
* HABP or VABP patients only: pulmonary disease that precludes evaluation of therapeutic response including known bronchial obstruction or a history of post-obstructive pneumonia, tracheobronchitis, primary lung cancer or malignancies metastatic to the lung, bronchiectasis, known or suspected active tuberculosis
* cUTI or AP patients only: renal abscess, chronic bacterial prostatitis, orchitis or epididymitis, polycystic kidney disease, one functional kidney, vesicoureteral reflux, renal transplant, cystectomy or ileal loop surgery, fungal UTI or complete, permanent obstruction of the urinary tract
* Patients in acute renal failure at the time of randomization
* Patients receiving intermittent hemodialysis (IHD) at the time of screening
* Pregnant or breastfeeding female patient

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-09-16 (Actual); Primary Completion 2016-08-18 (Actual); Study Completion 2016-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn E Connolly, MD, PhD, Study Director — Achaogen, Inc.

REFERENCES:
- [Derived] Kuti JL, Kim A, Cloutier DJ, Nicolau DP. Evaluation of Plazomicin, Tigecycline, and Meropenem Pharmacodynamic Exposure against Carbapenem-Resistant Enterobacteriaceae in Patients with Bloodstream Infection or Hospital-Acquired/Ventilator-Associated Pneumonia from the CARE Study (ACHN-490-007). Infect Dis Ther. 2019 Sep;8(3):383-396. doi: 10.1007/s40121-019-0251-4. Epub 2019 Jun 28. PMID 31254273

RESULTS

PARTICIPANT FLOW:
Groups:
- Plazomicin in Combination With Adjunctive Antibiotic: Cohort 2: Patients received 15 mg/kg as a 30 minute IV infusion once daily. Bloodstream infection (BSI), hospital acquired bacterial pneumonia (HABP), or ventilator associated bacterial pneumonia (VABP) patients received plazomicin and any supplemental antibiotic therapy, according to Investigator's choice, for 7 to 14 days. Complicated urinary tract infection (cUTI) or acute pyelonephritis (AP) patients received plazomicin monotherapy only for 4 to 7 days with an option to switch to oral therapy on or after Day 5.
Period: Overall Study
Arm/Group | Plazomicin in Combination With Meropenem or Tigecycline | Colistin in Combination With Meropenem or Tigecycline | Plazomicin in Combination With Adjunctive Antibiotic
Started | 18 | 21 | 30
Completed | 10 | 8 | 17
Not Completed | 8 | 13 | 13
Not completed — Death | 8 | 13 | 12
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population includes all randomized patients in Cohort 1 and all enrolled patients in Cohort 2.
Groups:
- Plazomicin in Combination With Meropenem or Tigecycline: Cohort 1: Patients received 15 mg/kg plazomicin therapy (plus meropenem or tigecycline) as a 30-minute IV infusion once daily for 7 to 14 days.
- Colistin in Combination With Meropenem or Tigecycline: Cohort 1: Patients received a 5 mg/kg IV loading dose (300 mg maximum) colistin (plus meropenem or tigecycline) followed by a 5 mg/kg/d maintenance dose divided into q8h or q12h for 7 to 14 days.
- Plazomicin in Combination With Adjunctive Antibiotic: Cohort 2: Patients received 15 mg/kg as a 30 minute IV infusion once daily. BSI, HABP, or VABP patients received plazomicin and any supplemental antibiotic therapy, according to Investigator's choice, for 7 to 14 days. cUTI or AP patients received plazomicin monotherapy only for 4 to 7 days with an option to switch to oral therapy on or after Day 5.
- Total: Total of all reporting groups
Arm/Group | Plazomicin in Combination With Meropenem or Tigecycline | Colistin in Combination With Meropenem or Tigecycline | Plazomicin in Combination With Adjunctive Antibiotic | Total
Number analyzed (Participants) | 18 | 21 | 30 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.94 (13.94) | 63.29 (18.25) | 62.8 (18.15) | 63.51 (16.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 7 | 24
  Male | 12 | 10 | 23 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16 | 17 | 29 | 62
  Black or African American | 1 | 1 | 0 | 2
  Asian | 1 | 0 | 0 | 1
  Multiple | 0 | 1 | 0 | 1
  Other Unspecified | 0 | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 0 | 8
  Not Hispanic or Latino | 13 | 18 | 29 | 60
  Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With All Cause Mortality (ACM) at Day 28 or Significant Disease-Related Complication (SDRC) in the Microbiological Modified Intent to Treat (mMITT) Population in Cohort 1
Description: ACM at Day 28: confirmed date of death within 28 days of the first dose of study drug, irrespective of causality. SDRCs for all patients: presence of 1 or more of the following complications within 7 days of randomization: new or worsening acute respiratory distress syndrome (ARDS), new lung abscess, new empyema, new onset of septic shock, new carbapenem-resistant Enterobacteriaceae (CRE) (HABP/VABP patients only); persistent bacteremia on study Day ≥5 (BSI patients only).
  Note: Although it is generally expected that results for primary and secondary endpoints will be presented for all arms included at baseline, results for Cohort 2 are not presented here as this Cohort was not part of the primary or key secondary endpoints per the protocol and statistical analysis plan (SAP).
Time Frame: Up to Day 28 for ACM, up to 7 Days for SDRCs in all patients, on or after Day 5 for BSI patients only.
Population: The mMITT population was a subset of the MITT population and included all patients who received ≥1 dose of study drug and had a CRE pathogen. CRE=meropenem minimum inhibitory concentration (MIC) of ≥4 micrograms per milliliter (μg/mL) or meropenem MIC=2 μg/mL and disk diffusion results (≤19 millimetres [mm]) indicating meropenem resistance.
Measure: Number; unit: percentage of patients
Arm/Group | Plazomicin in Combination With Meropenem or Tigecycline | Colistin in Combination With Meropenem or Tigecycline
Number analyzed (Participants) | 17 | 20
percentage of patients | 23.5 | 50
Statistical Analysis 1: Comparison: Plazomicin in Combination With Meropenem or Tigecycline vs Colistin in Combination With Meropenem or Tigecycline; Test type: Superiority — The 2-sided 90% confidence interval (CI) for the difference between groups in Cohort 1 (colistin minus plazomicin) is based on the unconditional exact method; 1-sided Fisher's exact test; Difference Estimate = 26.5, 90% CI 2-sided [-0.7 to 51.2]

2. Secondary Outcome: Percentage of Patients With ACM at Day 28 in the mMITT Population in Cohort 1
Description: ACM at Day 28: confirmed date of death within 28 days of the first dose of study drug, irrespective of causality.
  Note: Although it is generally expected that results for primary and secondary endpoints will be presented for all arms included at baseline, results for Cohort 2 are not presented here as this Cohort was not part of the primary or key secondary endpoints per the protocol and SAP.
Time Frame: Up to Day 28
Population: The mMITT population was a subset of MITT population and included all patients who received at least 1 dose of study drug and had a CRE pathogen. CRE=meropenem MIC of ≥4 μg/mL or meropenem MIC=2 μg/mL and disk diffusion results (≤19 mm) indicating meropenem resistance.
Measure: Number; unit: percentage of patients
Arm/Group | Plazomicin in Combination With Meropenem or Tigecycline | Colistin in Combination With Meropenem or Tigecycline
Number analyzed (Participants) | 17 | 20
percentage of patients | 11.8 | 40
Statistical Analysis 1: Comparison: Plazomicin in Combination With Meropenem or Tigecycline vs Colistin in Combination With Meropenem or Tigecycline; Test type: Superiority — [test comment as in outcome 1, analysis 1]; 1-sided Fisher's exact test; Difference Estimate = 28.2, 90% CI 2-sided [0.7 to 52.5]

3. Secondary Outcome: Percentage of Patients With Adjudicated Clinical Cure at the Test of Cure (TOC) Visit in the mMITT Population in Cohort 1
Description: Clinical response (CR) was assessed at end of treatment (EOT) in all patients and at TOC for those who were a clinical cure or had an indeterminate outcome at the most recent visit. Assessment of CR at TOC was not needed for those who were a clinical failure at an earlier visit. Clinical outcomes at both EOT and TOC were independently adjudicated by an external committee. The assessment was confounded by comorbidities and the occurrence of additional infections; thus, adjudicating CR of the baseline CRE infection was influenced by confounding signs and symptoms of unrelated infections or conditions. The difficulty assessing CR supports greater reliance on the more objective mortality-based primary endpoint in these patients.
  Note: Although it is generally expected that results for primary and secondary endpoints will be presented for all arms included at baseline, results for Cohort 2 are not presented here as this Cohort was not part of the endpoints per the protocol and SAP.
Time Frame: Up to TOC (Day 23)
Population: The mMITT population was a subset of MITT population and included all patients who received at least 1 dose of study drug and had a CRE pathogen. CRE=meropenem MIC of ≥4 μg/mL or meropenem MIC=2 μ/mL and disk diffusion results (≤19 mm) indicating meropenem resistance.
Measure: Number; unit: percentage of patients
Arm/Group | Plazomicin in Combination With Meropenem or Tigecycline | Colistin in Combination With Meropenem or Tigecycline
Number analyzed (Participants) | 17 | 20
percentage of patients
  EOT Visit: Clinical Cure | 64.7 | 45
  EOT Visit: Clinical Failure | 35.3 | 55
  TOC Visit: Clinical Cure | 35.3 | 35
  TOC Visit: Clinical Failure | 58.8 | 65
  TOC Visit: Indeterminate Response | 5.9 | 0
Statistical Analysis 1: Comparison: Plazomicin in Combination With Meropenem or Tigecycline vs Colistin in Combination With Meropenem or Tigecycline; Test type: Superiority — The 2-sided 90% confidence interval (CI) for the difference in clinical cure percentage at the TOC visit between groups in Cohort 1 (colistin minus plazomicin) is based on the unconditional exact method; 1-sided Fisher's exact test; Difference Estimate = -0.3, 90% CI 2-sided [-26.9 to 26.8]

4. Secondary Outcome: Time to Death Through Day 28 in the mMITT Population in Cohort 1
Description: Time to death through Day 28 is defined as days from first dose of study drug to death from any cause on or before Day 28. Patients who were alive at Day 28 were censored on Day 28. Any patient whose survival status was not known at Day 28 was censored on the last known date alive.
  Note: Although it is generally expected that results for primary and secondary endpoints will be presented for all arms included at baseline, results for Cohort 2 are not presented here as this Cohort was not part of the primary or key secondary endpoints per the protocol and SAP.
Time Frame: Up to Day 28
Population: The mMITT population included all patients who received at least 1 dose of study drug and had a CRE pathogen. CRE=meropenem MIC of ≥4 μg/mL or meropenem MIC=2 μg/mL and disk diffusion results (≤19 mm) indicating meropenem resistance.
Measure: Number; unit: percentage of patients
Arm/Group | Plazomicin in Combination With Meropenem or Tigecycline | Colistin in Combination With Meropenem or Tigecycline
Number analyzed (Participants) | 17 | 20
percentage of patients
  % of patients who died by Day 28 | 11.8 | 40.0
  % of patients censored at 28 days | 88.2 | 60.0
  % of patients censored at <28 days | 0.0 | 0.0
  Kaplan-Meier estmate of ACM at Day 28 | 11.8 | 40
Statistical Analysis 1: Comparison: Plazomicin in Combination With Meropenem or Tigecycline vs Colistin in Combination With Meropenem or Tigecycline; Test type: Superiority — The 2-sided 90% confidence interval (CI) for the unadjusted hazard ratio between groups in Cohort 1 (colistin:plazomicin) is based on a Cox proportional hazards regression model; 1-sided logrank test; Hazard Ratio (HR) = 3.97, 90% CI 2-sided [1.08 to 14.61]

5. Secondary Outcome: Percentage of Patients With ACM at Day 14 in the mMITT Population in Cohort 1
Description: ACM at Day 14 was defined as a confirmed date of death within 14 days of the first dose of study drug, irrespective of causality.
  Note: Although it is generally expected that results for primary and secondary endpoints will be presented for all arms included at baseline, results for Cohort 2 are not presented here as this Cohort was not part of the primary or key secondary endpoints per the protocol and SAP.
Time Frame: Day 14
Population: The mMITT population was a subset of MITT population and included all patients who received ≥1 dose of study drug and had a CRE pathogen. CRE=meropenem MIC of ≥4 μg/mL or meropenem MIC=2 μg/mL and disk diffusion results (≤19 mm) indicating meropenem resistance.
Measure: Number; unit: percentage of patients
Arm/Group | Plazomicin in Combination With Meropenem or Tigecycline | Colistin in Combination With Meropenem or Tigecycline
Number analyzed (Participants) | 17 | 20
percentage of patients | 5.9 | 20
Statistical Analysis 1: Comparison: Plazomicin in Combination With Meropenem or Tigecycline vs Colistin in Combination With Meropenem or Tigecycline; Test type: Superiority — The two-sided 90% confidence interval for the difference between groups in Cohort 1 (colistin minus plazomicin) is based on the unconditional exact method; 1-sided Fisher's exact test; Difference Estimate = 14.1, 90% CI 2-sided [-13 to 40.3]

6. Secondary Outcome: Percentage of Patients With Dose Adjustment Due to Therapeutic Drug Management (TDM)
Description: After the initial plazomicin dose, subsequent doses were adjusted, as directed, with the use of TDM on Day 1, 4, and 8 as needed.
  Note: Although it is generally expected that results for primary and secondary endpoints will be presented for all arms included at baseline, results for Cohort 1: Colistin are not presented here as TDM collection does not apply to and was not collected for patients in the colistin arm, as only plazomicin levels were measured.
Time Frame: Up to Day 14
Population: The safety population included all randomized patients who received any amount of study drug.
Measure: Number; unit: percentage of patients
Arm/Group | Plazomicin in Combination With Meropenem or Tigecycline | Plazomicin in Combination With Adjunctive Antibiotic
Number analyzed (Participants) | 18 | 30
percentage of patients | 77.8 | 86.7

7. Secondary Outcome: Percentage of Patients With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered to be drug related. An AE (also referred to as an adverse experience) can be any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, and it does not imply any judgment about causality. Adverse events also include the exacerbation or worsening of a condition present at screening other than the index infection for which the patient was enrolled in the study. A TEAE is any AE that newly appeared, increased in frequency, or worsened in severity following initiation of study drug. The safety population included all randomized patients who received any amount of study drug.
Time Frame: Up to Day 67
Population: The safety population included all randomized patients who received any amount of study drug.
Measure: Number; unit: percentage of patients
Arm/Group | Plazomicin in Combination With Meropenem or Tigecycline | Colistin in Combination With Meropenem or Tigecycline | Plazomicin in Combination With Adjunctive Antibiotic
Number analyzed (Participants) | 18 | 21 | 30
percentage of patients | 88.9 | 100 | 86.7

8. Secondary Outcome: Plasma Pharmacokinetics (PK): Area Under the Curve From 0 to 24 Hours (AUC 0-24h)
Description: PK specimens were collected on Days 1 and 4 using a sparse sampling scheme, and concentration-time data from these PK specimens were pooled with data from specimens collected for TDM. The pooled data were analyzed by population PK modeling, which described PK over the entire course of plazomicin treatment. The protocol allowed dose adjustments based on creatinine clearance; therefore, various dose regimens were used in the study, including regimens with dosing intervals of 12, 24, and 48 hours. To enable a combined summation of exposures across dose regimens, PK exposure parameters for the study were summarized for the first 48 hours of treatment. Thus, while exposures are summarized for the first 48 hours, the reported results considered patient data over the course of plazomicin treatment.
Time Frame: 48 hours
Population: PK population included all patients who had received at least 1 dose of plazomicin and had at least 1 quantifiable plazomicin plasma concentration available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/L (millgrams times hours per liter)
Groups:
- Plazomicin: All patients who received plazomicin throughout the study.
Arm/Group | Plazomicin
Number analyzed (Participants) | 48
mg*h/L (millgrams times hours per liter) | 235 (42)

9. Secondary Outcome: Plasma Pharmacokinetics (PK): Maximum Observed Plasma Drug Concentration (Cmax)
Description: as for outcome 8
Time Frame: 48 hours
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Plazomicin
Number analyzed (Participants) | 48
mg/L | 37.1 (39.3)

10. Secondary Outcome: Plasma Pharmacokinetics (PK): Minimum Observed Plasma Drug Concentration (Cmin)
Description: as for outcome 8
Time Frame: 48 hours
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Plazomicin
Number analyzed (Participants) | 48
mg/L | 2.1 (99.4)

ADVERSE EVENTS:
Time Frame: Up to Day 67
Description: The safety population included all randomized patients who received any amount of IV study drug. Because of the small sample size enrolled and the requirement to report AEs occurring in ≥5% of patients, all AEs are reported here, including those occurring in only a single patient.
Arm/Group | Plazomicin in Combination With Meropenem or Tigecycline | Colistin in Combination With Meropenem or Tigecycline | Plazomicin in Combination With Adjunctive Antibiotic
All-Cause Mortality (participants affected / at risk) | 8/18 | 13/21 | 12/30
Serious Adverse Events (participants affected / at risk) | 9/18 | 17/21 | 20/30
Other Adverse Events (participants affected / at risk) | 13/18 | 20/21 | 22/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Plazomicin in Combination With Meropenem or Tigecycline (N=18) | Colistin in Combination With Meropenem or Tigecycline (N=21) | Plazomicin in Combination With Adjunctive Antibiotic (N=30)
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0
Haemodynamic instability (Vascular disorders) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 2
Pneumonitis chemical (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 2 | 4
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 3 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Hyperosmolar state (Metabolism and nutrition disorders) | 0 | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0
Hepatitis infectious (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1
Pneumonia necrotising (Infections and infestations) | 0 | 0 | 1
Pseudomonal bacteraemia (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 3 | 0
Septic shock (Infections and infestations) | 4 | 5 | 5
Urinary tract infection (Infections and infestations) | 0 | 0 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Plazomicin in Combination With Meropenem or Tigecycline (N=18) | Colistin in Combination With Meropenem or Tigecycline (N=21) | Plazomicin in Combination With Adjunctive Antibiotic (N=30)
Hypotension (Vascular disorders) | 1 | 0 | 3
Pyrexia (General disorders) | 2 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 2 | 3
Depression (Psychiatric disorders) | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 2
Blood creatinine increased (Investigations) | 1 | 2 | 1
Blood fibrinogen decreased (Investigations) | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 2
Extrasystoles (Cardiac disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 3
Nausea (Gastrointestinal disorders) | 0 | 1 | 3
Vomiting (Gastrointestinal disorders) | 1 | 2 | 2
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 4 | 5
Renal impairment (Renal and urinary disorders) | 1 | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Penile ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Fungal sepsis (Infections and infestations) | 1 | 0 | 0
Oral fungal infection (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2 | 0
Sepsis (Infections and infestations) | 1 | 1 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0
Stoma site abscess (Infections and infestations) | 1 | 0 | 0
Systemic candida (Infections and infestations) | 1 | 0 | 0
Tinea cruris (Infections and infestations) | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator may publish/present the study results provided all of the following: (i) the primary publication has been published; or, if no such publication has occurred, at least 18m have passed since the completion of the study; (ii) Achaogen is allowed at least 60d to review; (iii) confidential information is deleted as requested; (iv) comments and proposed revisions are considered; and (v) during the 60d review, if requested, the Investigator shall delay the publication or presentation.